CLINICAL TRIAL: NCT02209376
Title: Pilot Study of Autologous T Cells Redirected to EGFRVIII-With a Chimeric Antigen Receptor in Patients With EGFRVIII+ Glioblastoma
Brief Title: Autologous T Cells Redirected to EGFRVIII-With a Chimeric Antigen Receptor in Patients With EGFRVIII+ Glioblastoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision to terminate prior to completion to pursue combination therapies.
Sponsor: University of Pennsylvania (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 35313, 820381
Record Dates: First submitted 2014-08-04; First posted 2014-08-05 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2019-03

CONDITIONS: Patients With Residual or Reccurent EGFRvIII+ Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Biological: CART-EGFRvIII T cells

INTERVENTIONS:
Biological: CART-EGFRvIII T cells

SUMMARY:
An Open-Label Phase 1 Pilot Study to determine the safety and feasibility of CART-EGFRvIII (autologous T cells transduced with a lentiviral vector to express a chimeric antigen receptor specific for EGFRvIII) in the treatment of patients with EGFRvIII+ glioblastoma who have had their first recurrence as determined by standard imaging or have have residual disease after initial resection.

ELIGIBILITY:
Inclusion Criteria:

* Pathological criteria: Glioblastoma (GBM) that is histologically confirmed by pathology review of surgically resected tissue.
* Tumor cells from resected tissue must be available for EGFRvIII testing. Patients who have previously been treated with an EGFRvIII-targeted therapy and recurred, must have a tumor sample obtained after their recurrence available for EGFRvIII testing.
* Age greater than 18 years.
* If the patient is on dexamethasone, the anticipated dose must be 4 mg/day or less for at least 5 days prior to apheresis.
* ECOG performance status of 0 or 1 Documented negative serum HCG for female patients of child-bearing potential.
* Participants with adequate organ function as measured by:

  * White blood count greater than or equal to 2500/mm^3; platelets greater than or equal to 100,000/mm^3, hemoglobin greater than or equal to 9.0 g/dL; without transfusion or growth factor support
  * AST, ALT, GGT, LDH, alkaline phosphatase within 2.5 x upper normal limit, and total bilirubin less than or equal to 2.0 mg/dL
  * Serum creatinine less than or equal to 1.5 x upper limit of normal
  * Coagulation tests PT and PTT have to be within normal limits, unless the patient has been therapeutically anti-coagulated for previous venous thrombosis.
* Provide voluntary informed consent for Tissue Screening and Apheresis

Inclusion Criteria Step 2:

1. Subject met all Step 1 Eligibility Criteria.
2. Tumor cells test positive for EGFRvIII expression (by RT-PCR, next generation sequencing, or immunohistochemistry) and a CART EGFRvIII product has been manufactured and formulated. Patients who have previously been treated with an EGFRvIII-targeted therapy and recurred are only eligible if a tumor sample obtained after their recurrence tests positive for EGFRvIII.
3. Stage of disease:

   * Cohort 1: Patients with first relapse of previously diagnosed primary glioblastoma. Recurrence may be determined by imaging and clinical criteria alone.
   * Cohort 2: Patients with newly diagnosed glioblastoma with a less than 95% resection or greater than or equal to 1 cm^3 of residual disease on the post-operative MRI (typically post-operative day 1).
4. If the patient is on dexamethasone, the dose must be 4 mg/day or less prior to CART-EGFRvIII infusion.
5. It is anticipated that all patients in Cohort 2 will have completed standard of care external beam radiotherapy and chemotherapy with temozolomide (TMZ) at the time of the pre-infusion safety visit.
6. Life expectancy less greater than 3 months
7. ECOG performance status of 0 or 1

9. Participants with adequate organ function as measured by:

* White blood count greater than or equal to 2500/mm^3; platelets greater than or equal to 100,000/mm^3, hemoglobin greater than or equal to 9.0 g/dL; without transfusion or growth factor support
* AST, ALT, GGT, LDH, alkaline phosphatase within 2.5 x upper normal limit, and total bilirubin less than or equal to 2.0 mg/dL
* Serum creatinine less than or equal to 1.5 x upper limit of normal
* Coagulation tests PT and PTT have to be within normal limits, unless the patient has been therapeutically anti-coagulated for previous venous thrombosis.
* Adequate cardiac function (greater than EF 55%) 10. Provide voluntary informed consent for study treatment. 11. Female subjects of reproductive potential must agree to use a reliable method of contraception.

Exclusion Criteria Step 1:

* Female subjects of reproductive potential who are pregnant or lactating. Female study participants of reproductive potential must have a negative serum pregnancy test as part of Step 1 eligibility confirmation.
* Uncontrolled active infection.
* Active or latent chronic hepatitis B [detectable hepatitis B surface antigen (HBsAg)] or active hepatitis C (positive serology [HCV Ab]) infection.
* HIV infection.
* Previous treatment with any gene therapy products.
* Known addiction to alcohol or illicit drugs.
* History of allergy or hypersensitivity to study product excipients (human serum albumin, DMSO, and Dextran 40)

Exclusion Criteria Step 2:

* Female subjects of reproductive potential who are pregnant or lactating. Female study participants of reproductive potential must have a negative serum pregnancy test within two weeks prior to CART-EGFRvIII cell infusion. The safety of this therapy on unborn children is not known.
* Uncontrolled active infection.
* Use of immunosuppressive agents such as cyclosporine, MMF, tacrolimus, or rapamycin within 4 weeks of enrollment on Step 2.
* A minimal dose of corticosteroid (dexamethasone up to 4 mg/day) is permitted. Recent or current use of inhaled steroids is not exclusionary.
* Previous treatment with any gene therapy products.
* Subjects or their physicians anticipate use of any of the following concurrent treatment or medications including: a. Radiosurgery (except for the Standard of Care Fractionated External Radiation therapy is a part of the protocol regimen in Cohort 2) b. Chemotherapy (except for the Standard of Care Temozolomide therapy in Cohort 2) c. Interferon (e.g. Intron-A®) d. Allergy desensitization injections e. Any ongoing investigational therapeutic medication. f. Bevacizumab
* Participants who have another cancer diagnosis with history of visceral metastases at the time of pre-entry evaluation. The following diagnoses are examples that will be allowed:

  * squamous cell cancer of the skin without known metastasis
  * basal cell cancer of the skin without known metastasis
  * carcinoma in situ of the breast (DCIS or LCIS)
  * carcinoma in situ of the cervix
  * prostate cancer with only PSA recurrence
  * any cancer that has not required systemic therapy (other than hormonal therapies) for the past three (3) years.
* Any uncontrolled active medical disorder that would preclude participation as outlined.
* Unstable angina and/or myocardial infarction within 6 months prior to screening
* Known addiction to alcohol or illicit drugs.
* History of allergy or hypersensitivity to study product excipients (human serum albumin, DMSO, and Dextran 40)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-11-18 (Actual); Primary Completion 2018-04-04 (Actual); Study Completion 2018-04-04 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Donald O'Rourke, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine; Susan Chang, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - UCSF, San Francisco, California
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Result] O'Rourke DM, Nasrallah MP, Desai A, Melenhorst JJ, Mansfield K, Morrissette JJD, Martinez-Lage M, Brem S, Maloney E, Shen A, Isaacs R, Mohan S, Plesa G, Lacey SF, Navenot JM, Zheng Z, Levine BL, Okada H, June CH, Brogdon JL, Maus MV. A single dose of peripherally infused EGFRvIII-directed CAR T cells mediates antigen loss and induces adaptive resistance in patients with recurrent glioblastoma. Sci Transl Med. 2017 Jul 19;9(399):eaaa0984. doi: 10.1126/scitranslmed.aaa0984. PMID 28724573
- [Derived] Tang OY, Tian L, Yoder T, Xu R, Kulikovskaya I, Gupta M, Melenhorst JJ, Lacey SF, O'Rourke DM, Binder ZA. PD1 Expression in EGFRvIII-Directed CAR T Cell Infusion Product for Glioblastoma Is Associated with Clinical Response. Front Immunol. 2022 May 6;13:872756. doi: 10.3389/fimmu.2022.872756. eCollection 2022. PMID 35603165
- [Derived] Yin Y, Boesteanu AC, Binder ZA, Xu C, Reid RA, Rodriguez JL, Cook DR, Thokala R, Blouch K, McGettigan-Croce B, Zhang L, Konradt C, Cogdill AP, Panjwani MK, Jiang S, Migliorini D, Dahmane N, Posey AD Jr, June CH, Mason NJ, Lin Z, O'Rourke DM, Johnson LA. Checkpoint Blockade Reverses Anergy in IL-13Ralpha2 Humanized scFv-Based CAR T Cells to Treat Murine and Canine Gliomas. Mol Ther Oncolytics. 2018 Aug 28;11:20-38. doi: 10.1016/j.omto.2018.08.002. eCollection 2018 Dec 21. PMID 30306125
- [Derived] Johnson LA, Scholler J, Ohkuri T, Kosaka A, Patel PR, McGettigan SE, Nace AK, Dentchev T, Thekkat P, Loew A, Boesteanu AC, Cogdill AP, Chen T, Fraietta JA, Kloss CC, Posey AD Jr, Engels B, Singh R, Ezell T, Idamakanti N, Ramones MH, Li N, Zhou L, Plesa G, Seykora JT, Okada H, June CH, Brogdon JL, Maus MV. Rational development and characterization of humanized anti-EGFR variant III chimeric antigen receptor T cells for glioblastoma. Sci Transl Med. 2015 Feb 18;7(275):275ra22. doi: 10.1126/scitranslmed.aaa4963. PMID 25696001